CLINICAL TRIAL: NCT04003727
Title: The Effect of Head Position on Glottic Visualisation and Intubation Success With Videolaryngoscope in Obese Patients
Brief Title: Glottic Visualisation During Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assoc. Prof., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 19-KAEK-085
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutral Position (Active Comparator): Head and neck will be on neutral position.
  Interventions: Device: Mcgrath Mac Videolaryngoscope
- Sniffing Position (Active Comparator): Head and neck will be on sniffing position
  Interventions: Device: Mcgrath Mac Videolaryngoscope
- Head Extension position (Active Comparator): Head will be on simple extension position
  Interventions: Device: Mcgrath Mac Videolaryngoscope

INTERVENTIONS:
Device: Mcgrath Mac Videolaryngoscope — Patient's laryngoscopy will be done using McGrath Mac video laryngoscope

SUMMARY:
In this study, we aimed to investigate the effects of head and neck positions on the visualization of glottis and the success of intubation during videolaryngoscopy in obese patients.

DETAILED DESCRIPTION:
Tree different head and neck positions will compare for glottic visualization and intubation success rates in obese patients (BMI> 30 kg / m2) who required endotracheal intubation for general anesthesia between 18-65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Being 18-65 aged
* Being obese
* Undergoing surgery under general anesthesia

Exclusion Criteria:

* Having difficult airway
* Being American Society of Anesthesiologist (ASA) 4 physical status
* Undergoing emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Glottic view | During laryngoscopy
  the percentage of glottic opening (POGO) and cormack-lehane scores will be used to rate of the glottic view
Intubation Success | During intubation
  Intubation attempt number will be recorded

SECONDARY OUTCOMES:
Intubation difficulty | During Laryngoscopy
  Intubation Difficulty Scale(IDS) score will be recorded.The IDS score is derived from seven variables. N1 represents the number of additional intubation attempts, N2 represents the number of additional operators, N3 is the number of alternative intubation techniques used; N4 represents the laryngoscopic view, N5 represents the lifting force applied during laryngoscopy, N6 represents the necessity to apply external laryngeal pressure to optimize glottic exposure, N7 represents the mobility of vocal cord. The IDS score is the sum of all variables and ranges from zero to infinity. A score of 0 indicates an easy tracheal intubation. Intubation is considered difficult if the score is greater than 5.
Intubation time | During Intubation
  The duration of the endotracheal tube placement will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karaman, MD, Principal Investigator — Tokat Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University Hospital, Tokat Province, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided